CLINICAL TRIAL: NCT02128178
Title: Laparoscopic Bariatric Surgery: Two Regimens of Venous Thromboprophylaxis: Prospective Randomized Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, MOHAMED ABDELLATIF, phd, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Enoxaparin
Record Dates: First submitted 2014-04-22; First posted 2014-05-01 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Morbid Obesity; Pulmonary Embolism
Keywords: Morbid obesity; Laparoscopic surgery; Compression ultrasonography; Pulmonary embolism; Bleeding
MeSH Terms: conditions — Obesity, Morbid; Pulmonary Embolism; Hemorrhage | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ENOXAPARIN 2 HOURS BEFORE (Active Comparator): Giving 40 mg enoxaparin SQ 2 hours before surgery and daily for 10 days thereafter
  Interventions: Drug: Enoxaparin 40 mg 2 hours before arm; Drug: Enoxaparin 40 mg 12 hours before arm
- Enoxaparin 40 mg 12 hours before (Active Comparator): Enoxaparin 40 mg 12 hours before surgery and once daily for 10 days thereafter
  Interventions: Drug: Enoxaparin 40 mg 2 hours before arm; Drug: Enoxaparin 40 mg 12 hours before arm

INTERVENTIONS:
Drug: Enoxaparin 40 mg 2 hours before arm — Enoxaparin 40 mg 2 hours before surgery
  Other Names: First group
Drug: Enoxaparin 40 mg 12 hours before arm — Enoxaparin 40 mg 12 hours before surgery
  Other Names: second group

SUMMARY:
Obese patients undergoing bariatric surgery warrant VTE prophylaxis because they are at high risk for developing a fatal pulmonary embolism or postthrombotic syndrome. However, a consensus does not exist on the most effective prophylactic approach.

DETAILED DESCRIPTION:
Two regimens of prophylaxis are supposed , the 1st one is to give enoxaparin 40mg 2 hours before surgery and continued daily for 10 days after, and the 2nd one is to start 12 hours before surgery and continued in the same way like the 1st one.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 OR >35 with comorbidities

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Venous thrombosis and/or pulmonary embolism (PE) | Postoperative 4 weeks
  To assess the venous thrombosis by compression ultrasonography and PE in suspected patients

SECONDARY OUTCOMES:
Bleeding from the surgery site , drain if any, GIT bleeding, | postoperative 4 weeks
  Bleeding from drain, GIT, or wounds are assessed clinically
hospital stay | 4 WEEKS
  hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: mohamed e abd ellatif, phd, Principal Investigator — Mansoura University
Locations (1):
- Manoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Amaral FC, Baptista-Silva JC, Nakano LC, Flumignan RL. Pharmacological interventions for preventing venous thromboembolism in people undergoing bariatric surgery. Cochrane Database Syst Rev. 2022 Nov 22;11(11):CD013683. doi: 10.1002/14651858.CD013683.pub2. PMID 36413425